CLINICAL TRIAL: NCT02468349
Title: IMproving reModeling in Acute myoCardial Infarction Using Live and Asynchronous TElemedicine.
Acronym: IMMACULATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Heart Centre, Singapore (Other)
Collaborators: National University of Singapore (Other); National University Hospital, Singapore (Other); Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Mark Chan, A/Prof Mark Chan, National University Heart Centre, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2014/00793
Record Dates: First submitted 2015-06-07; First posted 2015-06-10 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Left Ventricular Remodeling; Medication Adherence; Acute Coronary Syndrome
Keywords: Acute Myocardial Infarction; Telemedicine; Readmissions
MeSH Terms: conditions — Ventricular Remodeling; Medication Adherence; Acute Coronary Syndrome | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedicine (Experimental): The telehealth group will be remotely monitored and managed on medication adherence, dosage titration, and management of drug side effects, through a combination of feed-forward blood pressure monitoring, app-based education and medication reminders, and remote consultations.
  Interventions: Other: Telemedicine
- Standard care (No Intervention): The standard care group will receive face-to-face consultations at one month, 6 months and 12 months.

INTERVENTIONS:
Other: Telemedicine — Participants enrolled will be randomised 1:1 to either telemedicine arm or standard care arm.
  Arms: Telemedicine

SUMMARY:
The proposed research aims to compare Left ventricular remodeling outcomes among patients with AMI and elevated NT-pro-B-type natriuretic peptide receiving telemedicine-guided post-MI treatment vs. non-telemedicine guided treatment.

DETAILED DESCRIPTION:
Acute Myocardial Infarction (AMI) accounts for more than 6,000 admissions to Singapore hospitals each year. Contemporary treatment, including percutaneous intervention (angioplasty and stenting) and adjunctive drug therapy, has reduced early mortality from AMI.

In many healthcare systems, Hospital scorecards stipulate prescription of appropriate drugs upon discharge after hospitalization for AMI. These drugs include aspirin, a platelet P2Y12 inhibitor, angiotensin converting enzyme inhibitors (ACE-I) or angiotensin receptor blockers (ARB), beta-blockers and lipid-lowering drugs. Such quality improvement programs have led to an increase in prescription of these drugs upon discharge. Yet, 2 problems remain pervasive:

1. dose optimization; how the investigators escalate patients to the most effective drug doses, and
2. drug adherence; whether patients are taking these drugs regularly.

These 2 problems stem largely from the traditional model of episodic care entailing face-to-face visits between patient and healthcare practitioner. Inadequate dose optimization is most relevant to ACE-I/ARB and beta-blockers as healthcare practitioners necessarily prescribe low doses of these drugs at discharge to avoid excessive lowering of blood pressure soon after an AMI. Yet, these drugs are most effective at preventing adverse ventricular remodeling when patients take them at their maximum tolerated doses. In clinical trials, titrating these ACE-I/ARB and beta-blockers to target doses has required weekly outpatient visits, a model of care that most healthcare systems cannot afford.

The investigators hypothesize that a telemedicine-based system of care will lead to a greater reduction in ventricular remodeling as compared with usual care, by improving dose optimization and adherence to ACE-I/ARB and beta-blockers in patients with recent AMI.

Participants with AMI (n=300) will be recruited during the index hospitalization. A key inclusion criteria is an elevated NT-proBNP measurement during the index hospitalization. Participants will first undergo stratified randomization according to ST-segment classification (STEMI/NSTEMI), thereafter randomized into the Telehealth versus Control group in 1:1 sequential block randomization (blocks of 4 and 6). The telehealth intervention group will have their blood pressure and heart rate monitored twice daily at home for 2 months, with alternating titration between ACE-inhibitors and betablockers weekly during the first 2 months. After 2 months, they will continue on telemedicine consultation for 4 months; coaching on drug adherence, drug side-effects management and monitoring of symptoms. A smartphone-based app developed by PEACH Intellihealth will provide structured health education, medication reminders and real-time text messaging with telehealth professionals.

All participants enrolled will be put on 1 year of dual antiplatelet therapy, have a cardiac MRI done both at baseline and 6-months, and followed up with cardiologist review visit at 1, 6 and 12 months. Major adverse cardiovascular and cerebrovascular events will be assessed during each cardiologist review visit, and beyond 12 months, it will be assessed by either phone calls or online/mailed questionnaires at 18 and 24 months.

Four substudies have been planned: a substudy to assess the impact of telemedicine on readmissions (ALTRA), a substudy to assess the effect of telemedicine on adherence to antiplatelet therapy (TICA), a substudy to assess the cost-effectiveness of telemedicine (CEA) and a substudy to assess the effect of telemedicine on MR-PET measured cardiac work efficiency (CES).

ELIGIBILITY:
Inclusion criteria

1. Clinically diagnosed STEMI or NSTEMI* within the last 7 days at high risk of ventricular remodeling

   * Typical history of ischemic chest pain or angina equivalent symptoms (e.g. acute onset dyspnea)
   * Typical rise or fall of cardiac enzymes with at least one value of cardiac troponin I≥10 ug/L.
   * ECG changes required for diagnosis of STEMI: ≥0.1mV ST segment elevation in two or more contiguous limb leads or precordial leads or presence of Q waves ≥0.02 sec in two or more contiguous limb leads or precordial leads, or new onset left bundle branch block (LBBB), *The definition of STEMI and NSTEMI follows the 3rd universal definition of MI [19]
2. Pre-discharge NTproBNP ≥300 pg/mL for both STEMI and NSTEMI
3. Undergone PCI for the index event
4. Age >21 years and <85 years

Exclusion criteria

1. Hypersensitivity to ticagrelor, aspirin or any excipients
2. Active pathological bleeding
3. History of intracranial haemorrhage
4. Bacterial Infection within 6 weeks preceding the primary angioplasty, HIV, autoimmune disease (e.g. SLE, rheumatoid arthritis, scleroderma and Grave's disease, etc) or on immunosuppressive therapy
5. Women of child-bearing potential, known to be pregnant, breast-feeding, or intend to become pregnant during the study period
6. Malignancy within last 2 years
7. History of significant valvular heart disease (moderate or severe MS, MR, AS, AR, TR)
8. Planned CABG within the next 6 weeks
9. Unable to be weaned off inotropes or IABP
10. Active asthma or any other contraindications to beta-blockers
11. Arrhythmias precluding proper CMR image acquisition, such as atrial fibrillation and frequent atrial or ventricular ectopy of > 1 in 5 intrinsic QRS complexes
12. Contraindications to cardiac magnetic resonance imaging including claustrophobia, pacemaker or ICD implantation, mechanical valve or other metallic implants
13. Severe liver impairment due to chronic liver disease e.g. advanced alcoholic liver cirrhosis or primary biliary cirrhosis
14. Significant renal impairment (eGFR <50ml min-1), end stage renal failure on renal replacement therapy
15. Anaemia (Hb<10 g/dL).
16. Psychosocial barriers to telemedicine adoption (screening for education level, dementia, substance abuse and other psychological disorders)
17. Participants who cannot be followed up
18. Participants not able or willing to consent for study.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Difference in Left Ventricular End-Systolic Volume (ml) | 6 months
  Difference in Left Ventricular End-Systolic Volume (ml) measured on cardiac magnetic resonance imaging

SECONDARY OUTCOMES:
Haemodynamic Stress | 6 months
  Frequency of participants with reduction in NT-proBNP <20%
Infarct size (grams and % of total LV mass) | 6 months
  Infarct size (grams and % of total LV mass) measured on cardiac magnetic resonance imaging
Adenosine diphosphate-induced platelet reactivity | 6 months
  Difference in Multiplate ADP test (AU*min)
Hospitalisation & readmission | 2 years
  Difference in incidence of Death, MI, Stroke, readmission for recurrent ischaemia requiring unplanned revascularization and readmission for heart failure.

OTHER OUTCOMES:
Quality of Life | 2 years
  Difference in QoL outcome measures
Medication Adherence | 12 months
  Difference in medication adherence score and pill count

CONTACTS AND LOCATIONS:
Overall Officials: Mark Chan, Principal Investigator — National University Heart Centre, Singapore; A. Mark Richards, Study Chair — National University Heart Centre, Singapore
Locations (3):
- Singapore (3):
  - National Heart Centre Singapore, Singapore, National Heart Research Institute
  - National University Heart Centre Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnold SV, Spertus JA, Masoudi FA, Daugherty SL, Maddox TM, Li Y, Dodson JA, Chan PS. Beyond medication prescription as performance measures: optimal secondary prevention medication dosing after acute myocardial infarction. J Am Coll Cardiol. 2013 Nov 5;62(19):1791-801. doi: 10.1016/j.jacc.2013.04.102. Epub 2013 Aug 21. PMID 23973701
- [Derived] Chan MY, Koh KWL, Poh SC, Marchesseau S, Singh D, Han Y, Ng F, Lim E, Prabath JF, Lee CH, Sim HW, Chen R, Carvalho L, Tan SH, Loh JPY, Tan JWC, Kuwelker K, Amanullah RM, Chin CT, Yip JWL, Lee CY, Gan J, Lo CY, Ho HH, Hausenloy DJ, Tai BC, Richards AM; IMMACULATE Investigators. Remote Postdischarge Treatment of Patients With Acute Myocardial Infarction by Allied Health Care Practitioners vs Standard Care: The IMMACULATE Randomized Clinical Trial. JAMA Cardiol. 2021 Jul 1;6(7):830-835. doi: 10.1001/jamacardio.2020.6721. PMID 33377898